CLINICAL TRIAL: NCT00618319
Title: An Open-Label, 18FDG-PET Pharmacodynamic Assessment of the Effect of BIIB021 in Subjects With Gastrointestinal Stromal Tumors (GIST) Refractory to, Intolerant of, or Not a Candidate for Imatinib and Sunitinib Treatment
Brief Title: An Open-Label, 18FDG-PET Pharmacodynamic Assessment of the Effect of BIIB021 in Subjects With Gastrointestinal Stromal Tumors (GIST)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120GS201
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2011-03

CONDITIONS: GIST
MeSH Terms: interventions — 6-chloro-9-(4-methoxy-3,5-dimethylpyridin-2-ylmethyl)-9H-purin-2-ylamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): BIIB021
  Interventions: Drug: BIIB021

INTERVENTIONS:
Drug: BIIB021 — Dose, schedule, and duration specified in protocol
  Other Names: CNF2024

SUMMARY:
This study will examine the effect of BIIB021 on GIST growth and metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
* Age greater than or equal to 18 years at the time of informed consent.
* Pathologically confirmed GIST refractory to, intolerant of, or not a candidate for imatinib and sunitinib therapy.
* FDG PET standard uptake value (SUVmax; averaged over a maximum of 5 lesions) greater than or equal to 2 at screening.
* ECOG performance status of less than or equal to 2.
* Lab values consistent with adequate renal hepatic and bone marrow function.
* Must utilize effective contraception.

Exclusion Criteria:

* Prior treatment with imatinib, sunitinib, or sorafenib with in 14 days of day 1.
* Prior treatment with Hsp90 inhibitors at any time.
* Prior antitumor therapies including prior experimental agents, approved antitumor small molecules (excluding imatinib, sunitinib, or sorafenib) and biologics, or radiotherapy with in 28 days or <3 half lives (whichever is longer) before start of BIIB021treatment.
* Diabetes treated with insulin and/ or concurrent severe or uncontrolled other medical disease (i.e, systemic infection, hypertension, coronary artery disease, congestive heart failure).
* History of/ or predisposition to seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Changes in FDG-PET imaging | 28 days

SECONDARY OUTCOMES:
Characterize the safety profile of BIIB021 | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (3):
- United States (3):
  - Reseach Facility, Encinitas, California
  - Research Site, Santa Monica, California
  - Reseach Facility, San Antonio, Texas